CLINICAL TRIAL: NCT00495586
Title: Situations That do Not Require Antibiotics for Acute Exacerbations of Mild-to-moderate Chronic Obstructive Pulmonary Disease
Brief Title: Effectiveness of Antibiotic Therapy for Exacerbations of Chronic Obstructive Pulmonary Disease
Acronym: TRANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Carl Llor, Doctor, Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06/31
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Antibiotics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pills t.i.d. for 8 days
  Interventions: Drug: Placebo
- Amoxycillin and clavulanic acid (Active Comparator): Amoxycillin and clavulanate t.i.d. for 8 days
  Interventions: Drug: Amoxicillin and clavulanic acid

INTERVENTIONS:
Drug: Placebo — One pill to be taken every eight hours for 8 days
  Other Names: It's placebo
  Arms: Placebo
Drug: Amoxicillin and clavulanic acid — 500-125 mg to be taken every eight hours for 8 days
  Other Names: Augmentine 500-125 mg 24 pills
  Arms: Amoxycillin and clavulanic acid

SUMMARY:
The purpose of this study is to determine the effectiveness of antibiotic therapy for patients with acute exacerbations of mild-to-moderate chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Antibiotics are usually prescribed for acute exacerbations of chronic obstructive pulmonary disease (COPD) even though their benefit in mild-to-moderate COPD is not demonstrated. The aim of this study is to assess the effectiveness of antibiotic therapy for exacerbations of COPD, what clinical variables are associated with an improved clinical response with antibiotic therapy with respect to placebo and to identify which patients might recover from an acute exacerbation without antibiotic therapy. Methodology: prospective, randomised, double blind, placebo-controlled clinical trial, in which exacerbations (at least one criterion present: increase of dyspnoea, increase of sputum production and/or increase of purulence) of patients older than 40 yr., smokers or ex-smokers of more than 10 pack-years, with COPD and FEV1 greater than 50%, diagnosed by spirometry and a predicted ratio FEV1/FVC<0.7%. Exclusion criteria: severe COPD (FEV1<50%), active neoplasm, tracheotomy, pneumonia, hospitalization criteria, patients previously being on antibiotics, immunodepressed, history of hypersensitivity to beta-lactams or intolerance to clavulanate, enrollment in other clinical trials, patients who refuse to take part in this study, and patients who have not had a spirometry test for the past two years. Sample size: 677 patients. Interventions: first visit: the patient will be given details of the clinical trial and will be asked to sign informed consent; other data: sputum color, chest X-ray ordered to rule out pneumonia, C-reactive protein levels, and peak flow measurement. The patient will be randomised to receive amoxicillin plus clavulanate or placebo and will be scheduled to return for a 2nd follow-up visit after 3 or 4 days to assess the clinical response and peak flow measurements and to rule out any worsening of the condition. Third visit: scheduled after 9-11 days to assess the clinical response, drug-compliance and peak flow measurement. Fourth visit after 15-20 days for clinical assessment and to observe whether any relapses have occurred. Date of the following exacerbation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbations (at least one criterion present: increase of dyspnoea, increase of sputum production and/or increase of purulence) of
* patients older than 40 years old,
* smokers or ex-smokers of more than 10 pack-years,
* with COPD and FEV1 greater than 50%, diagnosed by spirometry and a predicted ratio FEV1/FVC<0.7%.

Exclusion Criteria:

* Severe COPD (FEV1<50%)
* Pneumonia
* Active neoplasm
* Tracheotomy
* Criteria for hospitalisation
* Patients previously being on antibiotics
* Immunodepressed patients
* History of hypersensitivity to beta-lactams or intolerance to clavulanate
* Enrollment in other clinical trials
* Patients who refuse to take part in this study
* Patients who have not had a spirometry test for the past two years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Llor, Doctor, Principal Investigator — Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC); Marc Miravitlles, Doctor, Study Director — Hospital Clinic; Ana Moragas, Family doc., Study Director — Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC)
Locations (13):
- Spain (13):
  - Hospital Clínic, Barcelona, Catalonia
  - Primary Healthcare Center La Marina, Barcelona, Catalonia
  - Primary Healthcare Center Figueres, Figueres, Catalonia
  - Primary Healthcare Center Montilivi, Girona, Catalonia
  - Primary Healthcare Center Girona-4, Girona, Catalonia
  - Primary Healthcare Centre Breda-Hostalric, Hostalric, Catalonia
  - Primary Healthcare Center Lleida, Lleida, Catalonia
  - Primary Healthcare Centre Molins de Rei, Molins de Rey, Catalonia
  - Primary Healthcare Centre Olot, Olot, Catalonia
  - Primary Healthcare Center Reus-3, Reus, Catalonia
  - Primary Healthcare Center Les Muralles, Tarragona, Catalonia
  - Primary Healthcare Centre Jaume I, Tarragona, Catalonia
  - Primary Healthcare Center Valls Urbà, Valls, Catalonia

REFERENCES:
- [Derived] Miravitlles M, Moragas A, Hernandez S, Bayona C, Llor C. Is it possible to identify exacerbations of mild to moderate COPD that do not require antibiotic treatment? Chest. 2013 Nov;144(5):1571-1577. doi: 10.1378/chest.13-0518. PMID 23807094
- [Derived] Llor C, Moragas A, Hernandez S, Bayona C, Miravitlles M. Efficacy of antibiotic therapy for acute exacerbations of mild to moderate chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Oct 15;186(8):716-23. doi: 10.1164/rccm.201206-0996OC. Epub 2012 Aug 23. PMID 22923662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 353 patients invited to participate in this trial, 32 did not fulfill the inclusion criteria (14 presented a forced expiratory volume in one second [FEV1]/forced vital capacity [FVC] ratio > 70% and 18 a FEV1<50%). Three more had a positive X-ray for pneumonia and were therefore excluded.
Period: Overall Study
Arm/Group | Placebo | Amoxycillin and Clavulanic Acid
Started | 156 | 162
Completed | 152 | 158
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Amoxycillin and Clavulanic Acid | Total
Number analyzed (Participants) | 156 | 162 | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 46 | 100
  >=65 years | 102 | 116 | 218
Age Continuous [Mean (Standard Deviation); unit: years] | 67.8 (11.0) | 68.4 (9.9) | 68.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 122 | 135 | 257
Region of Enrollment [Number; unit: participants]
  Spain | 156 | 162 | 318

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Were Cured
Description: Cure defined as the disappearance of the acute signs and symptoms related to the infection, with complete return to the previous situation of stability
Time Frame: Day 9-11
Population: Clinical cure at end of therapy visit at day 9-11 in the ITT population
Measure: Number; unit: Participants
Arm/Group | Placebo | Amoxycillin and Clavulanic Acid
Number analyzed (Participants) | 152 | 158
Participants | 91 | 117
Statistical Analysis 1: Comparison: Placebo vs Amoxycillin and Clavulanic Acid; For the comparison of the efficacy of antibiotic versus placebo, we accepted a null hypothesis if the cure rate in the intervention group was the same or ±7% as that observed in the placebo arm. Based on previous studies, the expected rate of cure among patients assigned to antibiotic therapy was 90%. For an alpha of 0.05 and a beta of 0.2 and accepting possible losses of 15%, we calculated that the sample size is 677 patients in total; Test type: Non-Inferiority or Equivalence — Equivalence; p < 0.05, Chi-squared; Mean Difference (Final Values) = 14.2, 95% CI 2-sided [3.7 to 24.3], Standard Deviation 9.5

2. Secondary Outcome: Number of Days Till the Next Exacerbation
Description: For the assessment of the time till next exacerbation patients were monitored over a period of 365 days on a three-monthly basis. Patients were instructed to contact their physician immediately if there was any change in their health status. Diagnosis of a new exacerbation was based on the same clinical criteria described previously. For the calculation of time to the next exacerbation, all clinical failures occurring during therapy were counted as zero exacerbation-free interval days.
Time Frame: One year
Population: Patients with clinical success at the end of therapy visit
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Amoxicillin and Clavulanic Acid: Eighty-three exacerbations were reported during the year of follow up among those patients who had clinical success at end of therapy visit (83/143: 58%)
- Placebo: Ninety exacerbations were reported during the year of follow up among those patients who had clinical success at end of therapy visit (90/123: 73.2%)
Arm/Group | Amoxicillin and Clavulanic Acid | Placebo
Number analyzed (Participants) | 143 | 90
Days | 233 [110 to 365] | 160 [66 to 365]

ADVERSE EVENTS:
Time Frame: 20 days
Arm/Group | Placebo | Amoxycillin and Clavulanic Acid
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/158
Other Adverse Events (participants affected / at risk) | 12/152 | 23/158
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=152) | Amoxycillin and Clavulanic Acid (N=158)
Gastrointestinal disturbance (Gastrointestinal disorders) | 9 (9) | 23 (23) — 32 cases
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The required sample size could not be achieved. This clinical trial was only partially funded by an independent academic institution without any other source of funding. However, due differences obtained the sample size allowed for a power of 80%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes